CLINICAL TRIAL: NCT07270211
Title: Magnetocardiography in Long QT Syndrome: A Prospective Study of Its Clinical and Prognostic Utility
Brief Title: MCG In Long QT Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mohamad Adnan Alkhouli, Principal Investigator, Mayo Clinic
Other Study IDs: 25-008283
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Magnetocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects diagnosed with atrial fibrillation
  Interventions: Diagnostic Test: Magnetocardiography

INTERVENTIONS:
Diagnostic Test: Magnetocardiography — MCG is a non-invasive, radiation-free imaging technique that detects the magnetic field generated by the electrical activity of the heart.

SUMMARY:
The primary objective of this observational study is to evaluate whether magnetocardiography (MCG) findings more accurately predict clinical outcomes in patients with acquired Long QT syndrome compared to ECG. The secondary objective is to assess differences in QT interval length between MCG and ECG. The primary safety objective is to characterize the safety profile of the CardiAQ MCG device.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years on the date of consent
2. Ability for participant to comply with study requirements
3. Written informed consent
4. Confirmed diagnosis of atrial fibrillation and receiving dofetilide for rhythm control in the inpatient setting.

Exclusion Criteria

1. Pregnant or breastfeeding
2. Active thoracic metal implants (including pacemaker, insertable cardiac monitor, or internal defibrillators).
3. External electrical pads or devices (e.g. Pacer pads, ECG electrodes, heart rate patch), that must remain on patient's chest during MCG scan
4. Inability to lie down in a supine/inclined position and stay still on the examination bed
5. Clinical conditions that in the opinion of the Investigator would compromise the safety of the patient or ability to complete the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study candidates may be identified and recruited in one of the following ways:
  * In-patient service at the study institution.
  * From the Principal Investigator or Co-Investigator clinical practices
  * Referral from other hospitals
  * Cardiology Specialty Clinics
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of successful dofetilide loading using Magnetocardiography | Baseline
  Dofetilide loading is considered successful if the following conditions are met:
  1. No excessive QTc prolongation QTc remains <500 ms, and no >15% increase from baseline.
  2. No sustained VT or recurrent/symptomatic non-sustained VT (NSVT) suggestive of proarrhythmia.
  3. No symptomatic bradycardia or hemodynamic instability
  4. Stable renal function
  5. No deterioration necessitating dose reduction or discontinuation.
  6. Discharge on a stable dose
Number of successful dofetilide loading using Electrocardiogram | Baseline
  Dofetilide loading is considered successful if the following conditions are met:
  1. No excessive QTc prolongation QTc remains <500 ms, and no >15% increase from baseline.
  2. No sustained VT or recurrent/symptomatic non-sustained VT (NSVT) suggestive of proarrhythmia.
  3. No symptomatic bradycardia or hemodynamic instability
  4. Stable renal function
  5. No deterioration necessitating dose reduction or discontinuation.
  6. Discharge on a stable dose

SECONDARY OUTCOMES:
Magnetocardiography - QT interval length | Baseline
  QT interval length is a measurement from the start of the Q wave to the end of the T wave. This will be measured in seconds.
Electrocardiogram - QT interval length | Baseline
  QT interval length is a measurement from the start of the Q wave to the end of the T wave. This will be measured in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Alkhouli, M.D., M.B.A., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No